CLINICAL TRIAL: NCT02094443
Title: A Multicenter, Open-label, Randomized, 2-arm, Phase II Trial of Pharmacodynamics, Pharmacokinetics and Safety of Two Dose Regimens of DEB025/Alisporivir in Combination With Ribavirin Therapy in Chronic Hepatitis C Genotype 2 and 3 Patients Who Have Previously Failed Interferon Therapy or Are Intolerant or Unable to Take Interferon.
Brief Title: Alisporivir With RBV in Chronic Hepatitis C Genotype 2 and 3 Participants for Whom Interferon is Not an Option
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDEB025A2233; 2013-003751-38 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Hepatitis C; Liver Disease
Keywords: Chronic hepatitis C genotype 2; Chronic hepatitis C genotype 3; Cyclophilin inhibitor; Interferon intolerant
MeSH Terms: conditions — Hepatitis C; Liver Diseases | interventions — alisporivir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alisporivir 300 mg BID (Experimental): Alisporivir (ALV) 300 mg twice daily (BID) with ribavirin for 12 or 24 weeks based on Week 2 response, with a safety follow-up of at least 4 weeks, during which patients did not receive any study medication
  Interventions: Drug: Alisporivir; Drug: Ribavirin
- Alisporivir 400 mg BID (Experimental): ALV 400 mg twice daily (BID) with ribavirin for 12 or 24 weeks based on Week 2 response, with a safety follow-up of at least 4 weeks, during which patients did not receive any study medication
  Interventions: Drug: Alisporivir; Drug: Ribavirin

INTERVENTIONS:
Drug: Alisporivir — ALV 100 and 200 mg soft gel capsules administered orally
  Other Names: DEB025
Drug: Ribavirin — RBV 200 mg tablets (weight-based dose: < 75 mg = 1000 mg/day; ≥ 75 kg = 1200 mg/day) administered orally in a divided daily dose
  Other Names: Copegus®

SUMMARY:
The primary purpose of this study is to evaluate the pharmacodynamic (i.e. hepatitis C virus (HCV) viral load), pharmacokinetic and safety profiles between two treatment groups receiving different doses of DEB025 in combination with ribavirin (RBV) during the first 12 weeks treatment in chronic hepatitis C genotype (GT)-2 and GT-3 patients who had previously failed interferon therapy or were intolerant or unable to take interferon.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed
2. Participants with HCV genotype 2 or 3 infection who have previously failed interferon therapy or are intolerant or unable to take interferon
3. Males or females aged ≥18 years
4. Diagnosed Chronic hepatitis C virus infection

Exclusion criteria:

1. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of that medication before enrollment
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
3. Hepatitis B surface antigen (HBsAg) positive
4. Human immunodeficiency virus (HIV) positive

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (9):
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Lancaster, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Seattle, Washington
- France (5):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris

RESULTS

PARTICIPANT FLOW:
Groups:
- Alisporivir 300 mg BID: Alisporivir (ALV) 300 mg twice per day (BID) with ribavirin (RBV) for up to 24 weeks.
- Alisporivir 400 mg BID: ALV 400 mg BID with RBV for up to 24 weeks.
Period: Overall Study
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Started | 26 | 26
Completed at Week 12 | 0 | 1
Completed at Week 24 | 11 | 8
Completed | 11 | 9
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Population: Full Analysis Set, defined as all participants who were correctly randomized.
Groups:
- Alisporivir 300 mg BID: ALV 300 mg BID with RBV for up to 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.25) | 54.5 (7.62) | 53.9 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatitis C Virus Ribonucleic Acid Viral Load at Week 12
Description: The change in log transformed Hepatitis-C Virus (HCV) Ribonucleic acid (RNA) from baseline to Week 12.
Time Frame: Baseline, Week 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
log10 IU/mL
  Baseline | 6.323 (0.4785) | 6.343 (0.6396)
  Change from baseline | -3.935 (2.3361) | -3.855 (2.7506)

2. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) at Week 12
Description: ALT levels were assessed as part of clinical chemistry assessments throughout the study as a measure of biochemical liver recovery. A negative change from baseline indicates less liver damage.
Time Frame: Baseline, Week 12
Population: Participants in the safety set with available data at the given time point
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 21 | 19
U/L
  Baseline | 77.3 (48.57) | 67.9 (42.94)
  Change from baseline | -67.4 (45.99) | -58.2 (44.50)

3. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response (SVR) 4, 12, and 24 Weeks After Treatment
Description: SVR is defined as HCV RNA less than the lower limit of quantification (LLOQ), i.e., <15 IU/mL, at 4 weeks (SVR4), 12 weeks (SVR12), and 24 weeks (SVR24) after treatment, respectively.
Time Frame: Up to 24 weeks posttreatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
percentage of participants
  SVR4 | 30.8 | 38.5
  SVR12 | 19.2 | 26.9
  SVR24 | 19.2 | 26.9

4. Secondary Outcome: Percentage of Participants With Extended Rapid Virologic Response
Description: Extended rapid virologic response (eRVR) was defined as serum HCV RNA < LLOQ after 2 weeks of treatment
Time Frame: 2 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
percentage of participants | 0.0 | 3.8

5. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: eRVR was defined as serum HCV RNA < LLOQ after 4 weeks of treatment
Time Frame: 4 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
percentage of participants | 3.8 | 15.4

6. Secondary Outcome: Percentage of Participants With End of Treatment Response (ETR)
Description: ETR was defined as serum HCV RNA < LLOQ at treatment end (completed or prematurely discontinued).
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
percentage of participants | 46.2 | 50.0

7. Secondary Outcome: Percentage of Participants With Abnormal Alanine Aminotransferase (ALT) at Baseline Who Had Normalized ALT at Treatment End and Study End
Description: ALT is an enzyme found mostly in the cells of the liver and kidney. When the liver is damaged, ALT is released into the blood. This makes ALT a common test for liver damage, because higher ALT levels may indicate more liver damage. ALT upper limit of normal is commonly considered to be 40 international units per liter (IU/L), so abnormal ALT is above 40 IU/L.
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Number analyzed (Participants) | 26 | 26
percentage of participants
  End of Treatment | 73.1 | 61.5
  End of Study | 38.5 | 42.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first subject first visit until last subject last visit. All reported serious adverse events occurred during treatment.
Description: The mean exposure to alisporivir and ribavirin or to their combination regimen was 17 weeks for the 300 mg arm and 15 weeks for the 400 mg arm.
Arm/Group | Alisporivir 300 mg BID | Alisporivir 400 mg BID
Serious Adverse Events (participants affected / at risk) | 3/26 | 3/26
Other Adverse Events (participants affected / at risk) | 22/26 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisporivir 300 mg BID (N=26) | Alisporivir 400 mg BID (N=26)
Coronary artery disease (Cardiac disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisporivir 300 mg BID (N=26) | Alisporivir 400 mg BID (N=26)
Hypertension (Vascular disorders) | 4 | 5
Fatigue (General disorders) | 6 | 6
Asthenia (General disorders) | 5 | 12
Anxiety (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 3
Irritability (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 4 | 4
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 4 | 7
Syncope (Nervous system disorders) | 2 | 2
Ocular icterus (Eye disorders) | 2 | 1
Dry eye (Eye disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritis generalised (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1
Bronchitis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other